CLINICAL TRIAL: NCT06739226
Title: Combination of CARTs, CTLs and DC Vaccines Targeting Melanoma
Brief Title: Combination Immunotherapy Targeting Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-24004
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: melanoma; CART; chimeric antigen receptor; CTL; DC; vaccine; GD2
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T/CTL/DCvac cells to treat melanoma (Experimental): Antigen-specific CAR T, CTL and DCvac to treat melanoma.
  Interventions: Biological: Antigen-specific CAR T, CTL and DCvac to treat melanoma.

INTERVENTIONS:
Biological: Antigen-specific CAR T, CTL and DCvac to treat melanoma. — Antigen-specific CAR T, CTL and DCvac to treat melanoma.

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of combination immunotherapy based on CAR T cells, cytotoxic T lymphocytes (CTLs), and dendritic cell (DC) vaccines modified with GM-CSF and B7-2 (CD86) against melanoma, which targets CAR T specific surface antigens such as GD2, CTL specific antigens such as MAGE-A4, gp100 and a pool of melanoma specific antigens presented by the DCs. Another goal of the study is to learn more about the function and persistence of the CAR T cells and antigen-specific immune effectors in patients.

DETAILED DESCRIPTION:
Melanoma, known for having the highest mutation burden among solid tumors, has seen a steady rise in incidence over recent years. Early-stage melanoma can often be treated by surgery. As the tumor invades deeper and cancer cells metastasize, the difficulty of radical surgery increases. Although targeted therapies have significantly improved survival rates for patients with advanced melanoma, the potential for drug resistance remains a significant challenge. In this context, immunotherapy has become a new area of exploration.Therapies such as chimeric antigen receptor (CAR) T cell therapy, cytotoxic T lymphocyte (CTL) therapy, and dendritic cell vaccines have demonstrated promising clinical outcomes across various tumor types. Moreover, clinical trials exploring the application of these immunotherapies for treating melanoma are advancing steadily. Consequently, this study aims to explore a novel approach to melanoma treatment by integrating these three distinct forms of immunotherapy.

CAR T cells are a specialized type of T cells engineered to recognize and eliminate tumor cells by targeting specific surface antigens. The selection of the appropriate target antigens is crucial for the efficacy of CAR T cell therapy. Recent research has identified several promising targets for melanoma treatment, including GD2, CD70, and CSPG4. The choice of target may depend on individual patient characteristics. Among these, GD2 is expressed on the surface of a majority of melanoma cells while being minimally present in normal tissues, making it a favorable target in melanoma treatment.

CTL therapy involves stimulating effector T cells with antigen-presenting cells targeting cancer-specific antigens. In order to enhance the tumor-specific immune response, these activated antigen-presenting cells are used to generate highly specific T cells. Studies have identified several melanoma-associated antigens, such as gp100, tyrosinase, Melan-A, MAGE-A1, MAGE-A4, and NY-ESO-1. gp100 and MAGE-A4 are expressed in a significant proportion of melanoma cells and are closely linked to the development and progression of the disease. Furthermore, aberrant expression of gp100 may be implicated in the malignant transformation of melanocytes.

The dendritic cell (DC) vaccine leverages DC to activate T cells that specifically recognize target antigens, with the goal of preventing cancer recurrence and controlling tumor growth. Research has shown that DC vaccines modified with immune modulators such as GM-CSF and B7-2 (CD86) hold potential for melanoma treatment. GM-CSF plays a critical role by upregulating the expression of Bcl-xL in DC cells and reducing their sensitivity to immunosuppressive cytokines, thereby ensuring the optimal function of DCs. B7-2 serves as a vital ligand for T cell activation. By modifying DCs with B7-2, the interaction between DCs and T cells is enhanced, and promoting T cell activation, which collectively contribute to anti-tumor response.

The primary objective of this study is to evaluate the feasibility, safety, and efficacy of a combination therapy that integrates CAR T cells, CTLs, and DC vaccines modified with GM-CSF and B7-2 (CD86) for the treatment of melanoma. Additionally, the study seeks to gain further insights into the function and persistence of CAR T cells and antigen-specific immune effector s in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with melanoma have received standard first-line therapy and have been diagnosed with non-resectable, metastatic, progressive or recurrent conditions.
* The expression of melanoma specific antigens is immunohistochemically stained and verified.
* Body weight greater than or equal to 40 kg.
* Age: ≥18 year and ≤ 75 years of age at the time of enrollment.
* Life expectancy: at least 8 weeks.
* Prior Therapy:

  1. There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must be resolved to grade 2 or less.
  2. Participants must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection.
  3. At least 7 days must have elapsed since the completion of therapy with any biologic agent, targeted agent, tyrosine kinase inhibitor or metronomic non-myelosuppressive regimen.
  4. At least 4 weeks must have elapsed since prior therapy that includes a monoclonal antibody.
  5. At least 1 week must has elapsed since any radiation therapy at the time of study entry.
* Karnofsky/jansky score of 70% or greater.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent.
* Pulse Ox greater than or equal to 90% on room air.
* Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
* Renal function: Patients must have serum creatinine less than 3 times ULN.
* Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable for hematologic toxicity.
* For all patients enrolled in this study, the patients or their legal guardians must sign an informed consent and assent.

Exclusion Criteria:

* Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, with the exception of grade 3 hematologic toxicity.
* Untreated central nervous system (CNS) metastasis: Patients with previous CNS tumor involvement that has been treated and is stable for at least 4 weeks following completion of therapy are eligible.
* Previous treatment with other genetically engineered CAR T cells.
* Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
* Patients who require systemic corticosteroid or other immunosuppressive therapy.
* Evidence of tumor potentially causing airway obstruction.
* Inability to comply with protocol requirements.
* Insufficient availability of T cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 1 year
  The toxicity profile of CAR T, CTL or DCvac is determined by Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Disease status is defined by the measurement of biochemical markers and image scan, and the outcome of treatment is classified as Complete Response/remission (CR), Very Good Partial Response/remission (VGPR), etc.
The expansion and persistency of antigen-specific CAR T cells | 1 year
  The investigators will monitor the expansion and functional persistency of CAR T cells in the peripheral blood of patients and examine their correlation with antitumor effects.
Immune responses after CAR T and CTL infusions and DCvac injections | 1 year
  IL-2 cytokine secretion profile will be assessed
Immune responses after CAR T and CTL infusions and DCvac injections | 1 year
  IFN-γ cytokine secretion profile will be assessed
Immune responses after CAR T and CTL infusions and DCvac injections | 1 year
  Anti-tumor effector activities will be assessed
Survival time of the patients | 3 years
  Progression free survival (PFS) of the patients treated with the CAR Ts, CTLs and DCvac will be evaluated.
Survival time of the patients | 3 years
  Overall survival (OS) of the patients treated with the CAR Ts, CTLs and DCvac will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No